CLINICAL TRIAL: NCT06377462
Title: Multicenter, Interdisciplinary National VEXAS Registry With Accompanying Biomaterial Collection
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Bristol-Myers Squibb (Industry); University Hospital Munich (Other)
Responsible Party: Sponsor
Other Study IDs: VEXAS-Registry
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: VEXAS Syndrome
Keywords: VEXAS
MeSH Terms: conditions — VEXAS syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 18 mL whole blood (peripheral venipuncture) and 9 ml bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is rapid collection of real-life data on the epidemiology, treatment and disease course in patients with VEXAS syndrome during routine clinical practice and collect biomaterials to evaluate genotype-phenotype associations, determine optimal treatment schedule, identify diagnostic features and biomarkers

DETAILED DESCRIPTION:
see brief summary

ELIGIBILITY:
Inclusion Criteria:

* Patients with established or suspected (clinical and hematological criteria) VEXAS Syndrome
* Age ≥18 years
* Signed informed consent form

Exclusion Criteria:

* patients who are not in a position to understand the nature and scope of participation in this register

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Planned recruitment: 20-30 patients/year
  * Number of planned study centres: 15-20
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of epidemiological data on VEXAS | enrollment
  incidence, age and sex distribution in adults in Germany
Collection and monitoring of initial disease manifestations | 5 years
  * spectrum and frequency of inflammatory manifestations
  * Association with hematological (pre)malignancies (MDS, Myeloma, MGUS, CHIP)
  * Monitor cardiovascular risk/thromboembolic events
Documentation of the treatment approaches and therapy sequences | 5 years
  Documentation of the treatment approaches and therapy sequences
Analysis of clinical-relevant clinical endpoints | 5 years
  complete remission (CR), hematological and clinical remission, molecular remissions, treatment-free remission (TFR)

SECONDARY OUTCOMES:
Describe disease cluster | 5 years
  * Phenotype cluster?
  * Genotype-phenotype associations?
  * Identification of biomarker?
Laboratory diagnostics | 5 years
  * Establish Diagnostic FACS signature
  * Establish biomarker for disease monitoring
  * Molecular characterization of the key regulatory gene UBA1, but also accompanying molecular mutations
  * Correlation with HLA polymorphisms
  * Coagulation Diagnostics
Correlation clinical endpoints with treatment approaches | 5 years
  Correlation clinical endpoints with treatment approaches
Quality of life data (QoL), fatigue questionnaire (Facit-F) | 5 years
  Quality of life data (QoL), fatigue questionnaire (Facit-F)
Accompanying translational research | 5 years
  * Metabolic signature
  * Inflammatory signature
  * Microbiome
  * Identify disease trigger /risc factors for disease onset
Collection of Biospecimens | 5 years
  Collection of Biospecimens

CONTACTS AND LOCATIONS:
Overall Officials: Katja Sockel, Dr. med., Study Chair — TU Dresden
Locations (13):
- Germany (13):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Evang. Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum rechts der Isar TUM, München
  - Klinikum Osnabrück GmbH, Osnabrück
  - Helios Kliniken Schwerin GmbH, Schwerin
  - Robert Bosch Gesellschaft für Medizinische Forschung mb, Stuttgart
  - Krankenhaus der Barmherzigen Brüder, Trier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website VEXAS Registry — https://vexas.net/